CLINICAL TRIAL: NCT07240090
Title: Relation of Craniovertebral Angle With Lumbar Proprioception and Trunk Muscles Strength in Patients With Cervical Radiculopathy
Brief Title: Relationship Between Craniovertebral Angle, Lumbar Proprioception, and Trunk Muscle Strength in Cervical Radiculopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Basma Ashraf Ali Mohamed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Basma Ashraf Ali Mohamed, Demonstrator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/005966; CU2025-01 (Other: Faculty of Physical Therapy ,Cairo University)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cervical Radiculopathy
Keywords: Craniovertebral Angle; Lumbar Proprioception; Trunk Muscle Strength; Cervical Radiculopathy; Forward Head Posture; Low Back Pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to

* Investigate the relation of cranio-vertebral angle with lumbar proprioception in patients with cervical radiculopathy.
* Investigate the relation of cranio-vertebral angle with trunk muscles strength in patients with cervical radiculopathy. Cervical radiculopathy is a condition that causes neck pain radiating to the arm due to nerve root compression. The study seeks to explore whether posture and trunk control are affected in these patients. Participants will be assessed for craniovertebral angle, lumbar proprioception, and trunk muscle strength using standardized physical therapy evaluation methods. The findings may help in understanding postural and neuromuscular changes associated with cervical radiculopathy and improve rehabilitation programs

DETAILED DESCRIPTION:
Cervical radiculopathy is a major disabling condition characterized by neck pain radiating to one or both of the upper extremities . Epidemiological data suggest that CR affects approximately 83 per 100,000 individuals annually, with peak incidence occurring between ages 40 and 50 years and a lifetime prevalence of 3.5% in the general population .

Cervical radiculopathy is a common neurological condition caused by nerve root compression. Cervical radiculopathy is frequently associated with neck pain and includes tingling, numbness, or discomfort in the arm, upper back, and upper chest with or without an associated headache. Frequent headaches, scapular pain, and sensory, motor and reflex dysfunction in the upper extremities are often associated with cervical radiculopathy. These symptoms can be extended to the neck muscles, zygapophyseal joints, intervertebral discs, nerve roots, or trunk. In addition, higher levels of self-reported disability are reported among patients with neck pain and cervical radiculopathy .

The underlying cervical spinal pathologies, including disc herniation, osteophyte formation, and spinal canal stenosis, are widely recognized as common precipitating factors for nerve root compression or inflammation in CR . Approximately 70-75% of CR cases co-occur with degenerative changes, while 20-25% are attributed to intervertebral disc herniation. Repetitive overloads and micro-injuries lead to spinal canal narrowing and disc degeneration via the hypertrophy of the spinal joints and the encroachment of surrounding structures. This degeneration promotes osteophyte formation, elevated levels of local prostaglandins causing inflammation near the dorsal root ganglion .

According to the latest Global Burden of Disease data, neck pain is the fourth leading cause of years lived with disability, following only back pain, major depressive disorder, and arthralgias .Over the past ten years, there has been an increase of 19% in both the prevalence of cervical spine pain and the number of years people have been disabled globally.

Forward head posture (FHP) is a poor habitual neck posture resulting from the prolonged inherence of a static awkward position .It is associated with muscle imbalance and joint decentration, particularly at the atlanto-occipital joint, C4-C5 segment, glenohumeral joint, cervicothoracic joint, and T4-T5 segment . FHP has been viewed as a cervical sagittal imbalance and is defined as an increase in C2-C7 sagittal vertical alignment (SVA). Lately, cervical sagittal vertical alignment has been found to be the most relevant parameter of cervical sagittal balance in distinguishing symptomatic subjects from asymptomatic subjects .

FHP-induced changes in cervical alignment exaggerate the extension of the upper cervical vertebrae (C1-C2) and flexion of the lower cervical vertebrae (C3-C7) in the sagittal plane, increasing the load on the cervical discs and joints . In FHP, the deep cervical flexor ,which plays an important role in the stability of the cervical vertebra, is weakened and elongated, resulting in lower cervical flexion, and the upper trapezius, suboccipital, semispinalis, splenius, sternocleidomastoid, and levator scapula muscles are shortened, resulting in hyperextension of the upper cervical vertebra . The occurrence of FHP is increasing as the time spent using smartphones and computers increases . FHP is also caused by carrying a heavy backpack, sitting in front of a computer screen for a long time without using a desk and chair properly for physique, and not exercising .

FHP evaluation is often based on the cranio-vertebral angle (CVA) between the horizontal line passing through the spinous process of C7 and the line connecting the tragus of the ear to the spinous process of C7 . The normal Craniovertebral angle ranges between 48-50 degrees, Anything less the 48 degrees is defined as Forward head . As CVA decreases, neck pain increases, leading to chronic pain that causes physical changes and dysfunction .

A forward head posture (FHP) produces various negative symptoms such as neck ache, shoulder pain, upper back pain, persistent headaches, increased curvature of the spine, and scapular dyskinesia . In the long run, this incorrect posture can injure not only the cervical vertebrae and ligaments but also the structures around the lumbar area .

Muscle imbalance due to long-term poor posture habits such as forward head posture leads to asymmetry and functional deterioration of the musculoskeletal system . In the past decade several publications have identified that head and neck alignment plays a role in whole body pain and impairment including LBP and related disorders. Studies have identified that several of the postural upright postural neurophysiological reflexes, are located within the head and neck region. Relatively few correlational studies were identified linking cervical spine alignment to thoracic spine ailments and full spine alignment to LBP it would seem logical that alterations in cervical spine alignment would influence, at least to some extent, pain and radiculopathy in lumbosacral disorders leading to low back pain .

Lower back pain (LBP) is a common musculoskeletal condition characterized by discomfort or pain in the lower region of the spine . Low back pain is a group of symptoms characterized by pain, muscle tension, soreness and/or stiffness from the bottom of the rib cage to the buttock folds, sometimes accompanied by sciatic pain . The lower back is the most commonly reported complaint area in musculoskeletal conditions, leading to pain, disability, and a reduction in overall life quality . LBP affects the physical, psychological, and social areas and carries a great socioeconomic burden, as it is the main cause of work absenteeism and the excessive use of therapeutic service.

Lumbar proprioception or Lumbar Repositioning Error (LRPE) refers to an individual's capacity to perceive and control the precise position of their lumbar spine. An adequate lumbar repositioning is crucial for sustaining spinal stability and an optimal function during activities. Proprioception involves conscious and unconscious awareness of joint position sense, kinesthesia, and force sense of body parts without vision, Since paraspinal muscles contain abundant muscle spindles ,they play an important role in generating proprioceptive signals to monitor midrange spinal motion . When lumbar repositioning is inaccurate, it can lead to ineffective movement patterns that might contribute to the development of low back pain.

Trunk muscles are the active neuromuscular system that responsible for maintaining stability of the spine as the spine needs to be mechanically stable at all times to avoid injuries that can eventually lead to pain. The trunk is the center of the kinematic chains, transferring forces and acting as a bridge between the upper and lower extremities. Multiple factors have been associated with the occurrence of LBP, among them the alteration of the neuromuscular response of the trunk . The deconditioning or decrease in the function of the lumbar musculature ,the reduction in the muscular mass of the trunk , and the reduction in the muscular strength of the trunk . Decreased trunk muscle strength could be considered risk factors for developing LBP, specifically isometric and isokinetic strength of trunk flexors and lumbar extensors muscles .

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical radiculopathy with ≥3 months history of neck pain radiating to only one upper extremity (unilateral)
* Patients with forward head posture and craniovertebral angle <50°
* Age between 30 and 55 years
* Body mass index (BMI) between 18 and 29.9 kg/m²

Exclusion Criteria:

* Cervical myelopathy
* Acute cervical radiculopathy
* Neck pain without radiculopathy
* Diabetic neuropathy
* Previous cervical surgery
* Cervical trauma
* Entrapment neuropathies in the upper limbs
* Rheumatoid arthritis
* Tumors or infections involving the cervical or lumbar spine
* Acute or chronic lumbar radiculopathy
* Vertebral fractures
* Lumbar spinal stenosis
* Cauda equina syndrome
* Previous lumbar surgery
* Lumbar spondylolisthesis

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 30-55 years diagnosed with cervical radiculopathy, of both sexes, attending outpatient clinics. Participants should be able to understand instructions to compete methods of assessment
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle | baseline
  The craniovertebral angle will be measured using digital photography to assess forward head posture in patients with cervical radiculopathy.
  The assessment of the FHP will be carried out by measuring the craniovertebral angle. Standing cervical posture alignment will be measured with photogrammetry, which provides a valid and reliable indicator of forward head posture using the CVA . A smartphone will be mounted on a tripod and positioned 1.5 meters away from the participant, with the height adjusted to the level of the participant's shoulder.
  Adhesive markers will be placed on a participant's C7 spinous process and tragus of the ear. The therapist will observe the participant from the lateral side while standing and then will take a picture of the participant from a fixed distance 1.5 meters
Tunk muscles strength | baseline
  Trunk flexor and extensor muscle strength will be measured once using an isokinetic dynamometer at two angular velocities (60°/s and 120°/s) to evaluate muscle performance in patients with cervical radiculopathy The Biodex System 3 Pro (Biodex Medical Systems IIVC;Shirley , Shirley, NY, USA) will be used to conduct the isokinetic and isometric trunk strength test . Peak torque will be the primary outcome to be asessed in trunk isokinetic variables, peak torque indicates the highest muscle force output through the range of motion and reflects muscle strength .The trunk range of movement will be limited at 50°, with 30° (-30°) of trunk flexion and 20° (+20°) of trunk extension. It will started from the flexion position and will be performed with 60°/s and 120°/s angular velocities
Lumbar proprioception | baseline
  Lumbar joint position sense will be assessed once by measuring the difference between the target and reproduced trunk flexion angle at 30 degrees using an isokinetic device to evaluate proprioceptive accuracy in patients with cervical radiculopathy The Biodex System 3 Pro Isokinetic Dynamometer (Biodex Medical Systems, Shirley, NY, USA) will be used to assess lumbar proprioception. The dynamometer with a specific reclining back attachment is designed to assess the lumbar region's repositioning accuracy. Its validity is ICC = 0.99 and reliability is ICC = 0.99 for evaluating joint position sensation. Testing active repositioning of the lumbar spine is at 30°/s During the training, the participants will be instructed to maintain a specific spinal range of motion, which range from neutral extension of the lumbar spine to 30° flexion. This range is chosen because of the ability of all participants to do it .

CONTACTS AND LOCATIONS:
Overall Officials: Rowida A Abdelgaleel, PhD, Study Director — Cairo University - Faculty of Physical Therapy
Locations (1):
- Faculty of Physical Therapy labs at Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Engebretsen KB, Taso M, Bjorland S, Jenssen HK, Skaara HE, Brox JI. A functional intervention within a cognitive approach to chronic cervical radiculopathy : Description of the non-surgical treatment arm in a randomised controlled trial evaluating the effectiveness of surgery. BMC Musculoskelet Disord. 2024 Aug 7;25(1):629. doi: 10.1186/s12891-024-07743-0. PMID 39112984
- [Background] Brea-Gomez B, Torres-Sanchez I, Ortiz-Rubio A, Calvache-Mateo A, Cabrera-Martos I, Lopez-Lopez L, Valenza MC. Virtual Reality in the Treatment of Adults with Chronic Low Back Pain: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Int J Environ Res Public Health. 2021 Nov 11;18(22):11806. doi: 10.3390/ijerph182211806. PMID 34831562
- [Background] Coleman M, Linieres J, Thery C, Gautier A, Daste C, Rannou F, Nguyen C, Lefevre-Colau MM, Roren A. Changes in isokinetic trunk muscle strength and endurance after two different restoration programs in people with chronic low back pain: A longitudinal retrospective study. Heliyon. 2024 Jul 20;10(15):e34914. doi: 10.1016/j.heliyon.2024.e34914. eCollection 2024 Aug 15. PMID 39145024
- [Background] Al-Shenqiti AM, Emara HA, Algarni FS, Khaled OA. Isokinetic trunk muscle performance in adolescents with different body mass indices. J Taibah Univ Med Sci. 2021 Apr 24;16(4):550-557. doi: 10.1016/j.jtumed.2021.03.008. eCollection 2021 Aug. PMID 34408612
- [Background] Alkhamees NH, Ali OI, Abdelraouf OR, Ibrahim ZM, Mohamed AA. Assessment of Isokinetic Trunk Muscle Strength and Fatigue Rate in Individuals after Bariatric Surgery. Medicina (Kaunas). 2024 Mar 26;60(4):534. doi: 10.3390/medicina60040534. PMID 38674180
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Baroncini A, Maffulli N, Al-Zyoud H, Bell A, Sevic A, Migliorini F. Nonopioid pharmacological management of acute low back pain: A level I of evidence systematic review. J Orthop Res. 2023 Aug;41(8):1781-1791. doi: 10.1002/jor.25508. Epub 2023 Feb 22. PMID 36811209
- [Background] Baroncini A, Maffulli N, Eschweiler J, Knobe M, Tingart M, Migliorini F. Management of facet joints osteoarthritis associated with chronic low back pain: A systematic review. Surgeon. 2021 Dec;19(6):e512-e518. doi: 10.1016/j.surge.2020.12.004. Epub 2021 Feb 10. PMID 33582054